CLINICAL TRIAL: NCT01574170
Title: Prospective Construction and Validation of a Prognostic Score to Identify Among Patients With Metastatic Breast Cancer Those Who Benefit From a Third Line Chemotherapy in Terms of Overall Survival
Acronym: METAL3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11 SEIN 07
Record Dates: First submitted 2012-03-16; First posted 2012-04-10 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Breast Cancer Starting a Third Line Chemotherapy
Keywords: Breast cancer,; Third line metastatic; Chemotherapy,; Overall survival,; Quality of life.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Construction of a prognostic score (non-drug intervention types) — Record of clinical, histological and biological data and questionnaires data in patients starting a third line metastatic until progression

SUMMARY:
This is a biomedical study of interventional type. The trial will include 270 patients (180 patients in the first cohort and 90 patients in a second cohort) over a period of 3 years + 2 years of follow up.

This prospective study will be conduct in patients who will receive a third line chemotherapy for metastatic breast cancer.

The main objective of the study (first cohort) is to identify patients who benefit from a third line treatment in terms of overall survival with a score established from clinical, histological, but also biological "classic" and "innovative" (account of circulating tumor cells) criteria, all of these criteria must be measurable before the introduction of the 3rd line.

This score will then be validated on the 2nd cohort.

There will be no interruption of inclusions between first and second cohort of patients

ELIGIBILITY:
Inclusion Criteria:

1. Women of more than 18 years old
2. WHO 0-4
3. Metastatic breast cancer
4. Progression after two lines of chemotherapy with treatment decision by investigator to start a third-line chemotherapy
5. Evaluable disease
6. Histology: breast carcinoma whatever the histological type, grade, hormone receptor expression and HER-2
7. Patient able to complete the EORTC PAL 15 Questionnaire
8. Patient member in a national insurance scheme
9. Informed consent obtained and signed by the patient

Exclusion Criteria:

1. History of other (s) cancer (s) potentially metastatic (s)
2. Woman participating in a third line chemotherapy clinical trial
3. Pregnant women or nursing mothers can not participate in the study
4. Patient under legal guardianship
5. Patient unable to undergo medical test for various reasons including social or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Overall survival defined as the time from patient inclusion to the date of death or date of last follow-up news (censured data) | 11 years

SECONDARY OUTCOMES:
The time to progression, defined as the time from patient inclusion to the date of the first documented tumor progression | 11 years
Quality of life using the EORTC QLQ-C15-PAL Questionnaire | 11 years
Patient satisfaction regarding therapeutic decisions at inclusion using a specific questionnaire developed by Llewellyn-Thomas | 11 years
Oncologists satisfaction regarding the management and communication with the patient will be studied at baseline and at the time or progression using the Likert ordinal scale | 7 years
Regret or not of the patient to have followed a 3rd line of chemotherapy will be recorded at the end of the treatment using the "Decision regret scale" Questionnaire, established by A. O'Connor | 11 years
Safety evaluated according to the classification of NCI CTCAE (Common Terminology Criteria for Adverse Events) V4.0 | 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence MD DALENC, Principal Investigator — Institut Claudius Regaud
Locations (16):
- France (16):
  - C.M.C.O. Claude Bernard, Albi
  - Institut de Cancérologie de l'Ouest Paul Papin, Angers
  - CHU Jean Minjoz, Besançon
  - CHRU Brest, Brest
  - Centre Hospitalier Jean Rougier, Cahors
  - Centre Hospitalier Intercommunal de Castres-Mazamet, Castres
  - Centre d'Oncologie et de Radiothérapie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier de Rodez, Rodez
  - Centre Paul Strauss, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - CHU Rangueil, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy